CLINICAL TRIAL: NCT06881771
Title: Investigating Genetic Causes and Molecular Mechanisms Responsible for Inherited Corneal Disease
Brief Title: FECD-TRACE: Fuchs' Endothelial Corneal Dystrophy TRAjectory and Correlation With Genotype in the United Kingdom
Acronym: FECD-TRACE
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 145682
Record Dates: First submitted 2025-02-28; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Fuchs Dystrophy; Fuchs' Endothelial Dystrophy; Fuchs' Endothelial Corneal Dystrophy of Bilateral Eyes; Corneal Dystrophy Fuchs; Corneal Dystrophy
Keywords: Fuchs' Corneal Endothelial Dystrophy; FECD; Corneal Dystrophies; Corneal Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Dystrophies, Hereditary; Corneal Dystrophy, Posterior Polymorphous, 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood-derived genomic DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-symptomatic FECD cohort: 1. Have at least one biological first-degree relative with a confirmed diagnosis of FECD AND have TCF4 gene CTG18.1 expansion ≥ 50 repeats OR
  2. Confirmed diagnosis of FECD by a qualified ophthalmologist but does not have clinically evident corneal oedema
  Interventions: Diagnostic Test: Clinical phenotyping; Genetic: CTG18.1 Expansion Status Genotyping
- Control cohort: 1. Have no known family history nor clinical features of FECD OR
  2. Have known family history of FECD but have been tested for the TCF4 gene CTG18.1 expansion and are not at genetic risk for FECD (CTG < 50 repeats).
  Interventions: Diagnostic Test: Clinical phenotyping; Genetic: CTG18.1 Expansion Status Genotyping

INTERVENTIONS:
Diagnostic Test: Clinical phenotyping — * Visual acuity assessment
  * Contrast sensitivity evaluation
  * Slit-lamp photography
  * Specular microscopy
  * Scheimpflug tomography
  * Anterior segment optical coherence tomography
  * In vivo confocal microscopy
  * Spatio-temporal optical coherence tomography
Genetic: CTG18.1 Expansion Status Genotyping — Genotyping for trinucleotide repeat in the TCF4 gene (CTG18.1) and other genetic biomarkers using blood or saliva derived genomic DNA. This includes:
  * Short tandem repeat - PCR
  * Triplet-repeat primed - PCR
  * Genome-wide single nucleotide polymorphism genotyping
  * Ultra-deep locus-specific next-generation sequencing

SUMMARY:
FECD-TRACE is an integral component of a large research program dedicated to Fuchs Endothelial Corneal Dystrophy (FECD) in the United Kingdom. This longitudinal, observational study aims to comprehensively characterize a cohort of younger research participants who have a genetic predisposition to developing FECD. By utilizing advanced anterior segment imaging techniques, the study will monitor these individuals over a span of several years, capturing phenotypic changes that reflect the progression of the disease. Concurrently, genetic biomarkers will be examined to establish correlations with the observed phenotypic changes. The primary objective of FECD-TRACE is to enhance our understanding of the intricate genetic mechanisms underlying FECD and establish connections between these genetic findings and clinical outcomes. Ultimately, this research strives to facilitate the development of personalized care approaches for individuals affected by FECD.

DETAILED DESCRIPTION:
FECD is the most prevalent repeat expansion disease in humans. Clinical anticipation and intergenerational expansion of disease-associated repeats are features of other repeat expansion diseases, but this area has not been comprehensively addressed in FECD. Due to its insidious onset and slow disease progression, early diagnosis of FECD in pre-symptomatic patients is challenging.

To gain insights into the variable penetrance of FECD and to identify early signs of the disease in genetically predisposed but asymptomatic individuals (i.e., a pre-symptomatic cohort), we aim to recruit biological relatives of FECD patients receiving care at study sites, as well as individuals with early-stage disease. By combining genotyping and clinical phenotyping, we seek to elucidate the underlying factors influencing disease manifestation.

Our deep phenotyping approach encompasses an array of advanced imaging techniques such as visual acuity assessment, contrast sensitivity evaluation, slit-lamp photography, specular microscopy, Scheimpflug tomography, and anterior segment optical coherence tomography. These cutting-edge modalities enable the detection of subclinical corneal edema by revealing subtle changes in corneal shape, volume, and reflectivity at a high resolution.

The imaging data obtained from participants will undergo meticulous quantitative analysis, allowing for the classification of anterior segment features and extraction of image-derived phenotypes. To capture the dynamic nature of FECD, eligible participants will be invited for follow-up examinations, facilitating a longitudinal assessment of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent for participation in the study
* Willing to attend scheduled study visits and undergo a clinical examination
* Willing to donate blood/saliva samples
* Fulfil the abovementioned cohort criteria

Exclusion Criteria:

* Presence of a secondary cause for corneal endothelial dysfunction or oedema
* Presence of clinically evident corneal oedema
* History of concurrent corneal diseases
* History of corneal surgeries, including corneal transplantation
* Cognitive impairment or inability to provide informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants meeting the recruitment criteria across multiple sites will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial cell density measurement (cells/mm2) | Baseline
  Specular Microscopy - Endothelial cell density.
CTG18.1 allele length (in number) | Baseline
  Polymerase Chain Reaction (PCR) will be performed from DNA (blood sample)
Detection of guttata (cells/mm2) | Baseline
  In Vivo Confocal Microscopy (IVCM) - Detection of guttata
Corneal thickness (in micrometers) | Baseline
  Anterior Segment Optical Coherence Tomography (AS-OCT) - Corneal thickness
Documentation of early corneal guttata development (Binary) | Baseline
  Slit-Lamp Photography - Documentation of early corneal guttata development.
Best-corrected visual acuity in LogMAR scale | Baseline
  Visual acuity measured by LogMAR chart
Corneal nerve density (nerves/mm2) | Baseline
  In Vivo Confocal Microscopy (IVCM) - Detection of nerves

CONTACTS AND LOCATIONS:
Overall Officials: Alice Davidson, PhD, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided